CLINICAL TRIAL: NCT04999241
Title: The Role of Combined Application of Exclusive Enteral Nutrition in the Induction of Remission for Children With Newly Diagnosed Moderate to Severe Ulcerative Colitis
Brief Title: Combined Application of EEN in the Induction of Remission in PUC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Chief of Gastroenterology, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC1.2
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Exclusive Enteral Nutrition; Ulcerative Colitis; Children
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adrenal Cortex Hormones; Infliximab; Mesalamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEN combined therapy group (Experimental): in the induction of remission phase, EEN will be used combine with corticosteroids or infliximab
  Interventions: Combination Product: exclusive enteral nutrition
- Non EEN combination group (Active Comparator): in the induction of remission phase, corticosteroids or infliximab will be used without EEN
  Interventions: Combination Product: regular food

INTERVENTIONS:
Combination Product: exclusive enteral nutrition — Administration of a liquid formula diet with the exclusion of all other regular food for 8 weeks, then patients can administration of regular food.
  Other Names: corticosteroids, infliximab, 5-ASA, AZA
  Arms: EEN combined therapy group
Combination Product: regular food — Administration of regular food in the induction phase and the later time.
  Other Names: corticosteroids, infliximab, 5-ASA, AZA
  Arms: Non EEN combination group

SUMMARY:
The role of exclusive enteral nutrition (EEN) in the induction of remission in pediatric patients with Crohn's disease had been well documented. But the role of EEN in children with Ulcerative Colitis (UC) was not clear. In this study, EEN will be combined with corticosteroids or infliximab in the induction of remission in pediatric UC patients with moderate to severe disease activity. The mucosal healing rate at week12 will be compared between the two groups (combine with EEN group VS non-combine group).

DETAILED DESCRIPTION:
The role of exclusive enteral nutrition (EEN) in the induction of remission in pediatric patients with Crohn's disease(CD) had been well documented. Several randomized controlled trial studies found that the overall induction of remission was equipotent with EEN compared to corticosteroids for pediatric CD. However, in promoting mucosal healing and improving the nutritional status, EEN was much better than corticosteroids. But the role of EEN in children with Ulcerative Colitis (UC) was not clear. In this study, EEN will be combined with corticosteroids or infliximab in the induction of remission in pediatric UC patients with moderate to severe disease activity. The mucosal healing rate at week 12 will be compared between the two groups (combine with EEN group VS non-combine group).The sustained corticosteroid-free clinical remission rate and treatment modification rate during the first year will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed UC
2. Years 6 to 18
3. Moderate to severe disease activity at diagnosis

Exclusion Criteria:

1. With mild disease activity at diagnosis
2. Had been treated with corticosteroids or biologics

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The mucosal healing rate | 12 week after intervention
  The Ulcerative Colitis Endoscopic Index of Severity (UCEIS) ≦1 points is defined as mucosal healing. This will be evaluated by inflammatory bowel disease endoscopist.

SECONDARY OUTCOMES:
sustained corticosteroid-free clinical remission rate | 1 year after intervention
  Sustained pediatric Ulcerative Colitis activity index (PUCAI) score <10 points during follow-up (week 14 to week 54 after intervention) without the treatment of corticosteroids . This will be evaluated by gastroenterologist.
Treatment modification rate | 1 year after intervention
  The rate of new treatment measures needed to be started due to worsening of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, Study Director — Children's Hospital of Fudan University